CLINICAL TRIAL: NCT05770908
Title: Web Application Based on Multimedia Animations to Support Therapeutic Exercise for Rotator Cuff Related Shoulder Pain: a Randomized Controlled Trial
Brief Title: Multimedia Animations to Support Therapeutic Exercise for Rotator Cuff Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Union (Other)
Responsible Party: Principal Investigator, Irene Pérez Porta, Principal Investigator, Hospital Universitario Fundación Alcorcón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI18/16
Record Dates: First submitted 2023-03-03; First posted 2023-03-16 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Impingement Syndrome; Rotator Cuff Tendinitis; Rotator Cuff Related Shoulder Pain
Keywords: Rotator Cuff Related Shoulder Pain; Therapeutic Exercise; Web-based video
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigators involved in the recruitment, and data analysis will be masked of participant's allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia animation videos plus paper-based therapeutic exercise program (Experimental)
  Interventions: Other: Therapeutic exercise program; Other: Multimedia animation information; Other: Paper-based information
- Paper-based therapeutic exercise program (Active Comparator)
  Interventions: Other: Therapeutic exercise program; Other: Paper-based information

INTERVENTIONS:
Other: Therapeutic exercise program — Therapeutic exercise program based on increasing resistance with elastic bands or weights. The programmes are composed of combinations of the following exercises:
  * Scaption with elastic band.
  * External rotation at 0º of abduction with elastic band.
  * Internal rotation at 0º of abduction with elastic band.
  * Shoulder protraction in supine position with weights.
  * Low row with elastic band.
  * Horizontal adduction stretching.
Other: Multimedia animation information — Multimedia animation videos (including audio) showing the performance of the prescribed exercises.
  Arms: Multimedia animation videos plus paper-based therapeutic exercise program
Other: Paper-based information — Paper-based information showing the performance of the prescribed exercises, based on figures and a brief description of the exercise performance.

SUMMARY:
The goal of this randomized controlled trial is to evaluate the benefits from adding multimedia animations to a paper-based therapeutic exercise program in subjects with rotator cuff related shoulder pain. The main question[s] it aims to answer are:

* Does subjects improve more regarding shoulder disability and pain?
* Are the subjects more satisfied with the treatment received?
* Do the subjects adhere more to the exercise program?
* Do the subjects have greater expectations with the treatment received? Participants will perform a therapeutic exercise program within 6 months. Researchers will compare the addition of web-app animations to the classical paper-based information.

ELIGIBILITY:
Inclusion Criteria:

* Presence of rotator cuff related shoulder pain, diagnosed as unilateral shoulder pain, located in the anterior and/or lateral deltoid region, which is reproduced by active elevation and/or lying on ipsilateral side, and with at least one the following orthopaedic tests: Neer, Hawkins-Kennedy and/or empty can.
* Pain lasting from at least 3-months.
* Pain intensity at rest, during movement, and sleeping ≥ 3/10 points on a numeric pain rating scale.
* To have a mobile phone, tablet or computer with internet connection.
* To understand written and spoken Spanish language.

Exclusion Criteria:

* History of major trauma or surgery on the shoulder, elbow, or cervical spine.
* Signs of other shoulder pathologies such as instability, frozen shoulder, calcific tendonitis, severe arthrosis, or neuralgic amyotrophy.
* Presence of full-thickness rotator cuff tears on ultrasound imaging.
* Signs and/or symptoms of neck-related shoulder pain and/or radiculopathy or radicular pain.
* Systemic diseases such as cancer, rheumatic disorders, sclerosis multiple, neurological disorders, etc.
* Severe psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) | Change from baseline to 6-week, change from baseline to 12-week, and change from baseline to 24-week
  The SPADI ranges from 0% (no disability) to 100% (maximum degree of disability)

SECONDARY OUTCOMES:
Change in Pain intensity | Change from baseline to 6-week, change from baseline to 12-week, and change from baseline to 24-week
  Mean pain intensity during last week (at rest, with movement, and at night) measured with a numeric pain rating scale, which ranges from zero (no pain) to 10 (worst pain imaginable).
Change in Patient's expectations of improvement | Change from baseline to 3-week, and change from baseline to 6-week
  Patient's expectations of improvement measured with a numeric rating scale, which ranges from 0 (no expectation of improvement) to 10 (full recovery expectation).
Patient's satisfaction | 6-week, and 12-week
  Patient's satisfaction with received treatment measured with a numeric rating scale, which ranges from zero (not at all satisfied with the treatment received) to 10 (fully satisfied with the treatment received)
Patient's impression of improvement | 6-week, 12-week, and 24-week
  Patient's impression of improvement measured with the Patient Global Impression of Improvement (PGI-I) scale. The PGI-I is an seven-point ordinal scale ranging from 1 (much worse), through 3 (no change), to 6 (very much better).
Patient's perceived usability of multimedia animations | 12-week
  Patient's perceptions on the usability of the multimedia animations measured with the System Usability Scale (SUS), which is composed of 10 items that are rated in a 5-point Likert-type scale from 1 (strongly disagree) to 5 (strongly agree), with an overall rating ranging from 0% of perceived usability to 100% of perceived usability.
Patient's perceived usefulness of multimedia animations | 12-week
  Patient's perceived usefulness of multimedia animations measured with a 5-point Likert-type scale, which ranges from 1 (strongly disagree) to 5 (strongly agree).
Patient's satisfaction with the multimedia animations | 12-week
  Patient's satisfaction with the multimedia animations measured with a 5-point Likert-type scale, which ranges from 1 (strongly disagree) to 5 (strongly agree).
Patient's adherence | 3-week, 6-week, 12-week, and 24-week
  Patient's home adherence to the prescribed exercises measured with self-registered calendars, as the percentage of days performing the exercise at home over the maximum days available between the first physical therapy session and the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Porta I, Florez-Garcia MT, Garcia-Perez F, Fernandez-Matias R, Perez-Manzanero MA, Araujo-Narvaez AM, Urraca-Gesto MA, Fernandez-Lagarejos C, Plaza-Manzano G, Perez-Fernandez E, Velasco-Arribas M. Effects of a web application based on multimedia animations to support therapeutic exercise for rotator cuff-related shoulder pain: protocol for an open-label randomised controlled trial. BMJ Open. 2024 Jul 22;14(7):e085381. doi: 10.1136/bmjopen-2024-085381. PMID 39038866